CLINICAL TRIAL: NCT03875885
Title: CONNECTing Caregivers to Supportive Services (CONNECT): A Technology-Based Intervention to Connect Cancer Caregivers With Supportive Care Resources
Brief Title: CONNECTing Head and Neck Caregivers to Supportive Care Resources
Acronym: CONNECT-HNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00056635; 5KL2TR001421-04 (NIH); WFBCCC 99519 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2019-03-04; First posted 2019-03-15 (Actual); Results first posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer Caregivers
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONNECT Intervention Group - Group A (Other): A web-based intervention (CONNECT) to empower and connect caregivers of newly diagnosed cancer patients to supportive care resources A randomized pilot study will be conducted to assess feasibility and acceptability and obtain data on caregiver and patient outcomes. CONNECT e-tool, re-education and optional referral (2 weeks post CONNECT e-tool). Baseline, one month post randomization data collection, three months post randomization data collection, quantitative and qualitative measures.
  Interventions: Behavioral: CONNECT
- CONNECT Comparison Group - Group B (Other): Baseline, one month post randomization data collection, three months post randomization data collection, quantitative and qualitative measures.
  Interventions: Behavioral: CONTROL

INTERVENTIONS:
Behavioral: CONNECT — A novel web-based intervention with input from an advisory panel of cancer caregivers, oncology providers, and psychosocial oncology professionals empowering caregivers with needs to seek services by providing education about the benefits of supportive care resources, systematically identifying their unmet needs, and connecting them with tailored supportive care resources.
  Arms: CONNECT Intervention Group - Group A
Behavioral: CONTROL — This group will receive a generic resource list. The generic resource list will be printed for participants and emailed to them, if participants have an email address.
  Arms: CONNECT Comparison Group - Group B

SUMMARY:
The purpose of this research is to determine feasibility and acceptability of randomized pilot trial to evaluate a technology-based intervention (CONNECT) to empower and educate caregivers about the benefits of supportive care resources, identify their unmet needs, and connect them with resources.

DETAILED DESCRIPTION:
The registration is for Objective two and three that refers to the clinical trial. The investigators will determine their ability to recruit caregivers of patients with head and neck cancer being treated at Wake Forest Baptist Comprehensive Cancer Center to a study that uses a technology-based intervention, CONNECT, which may increase head and neck cancer caregivers' knowledge about the benefits of supportive care resources, identify their unmet needs, and connect them with supportive care resources. In this study the investigators also want to look at their ability to recruit a control group of caregivers, that is, caregivers of patients with head and neck cancer being treated at Wake Forest Baptist Comprehensive Cancer Center that will receive a list of supportive care resources. Control groups are used in research to see if the intervention being studied really does have an effect. In addition, the investigators will determine whether or not the intervention has led to improvements in caregivers' use of supportive care resources, quality of care, and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

Eligible caregivers include those who are:

* Caregivers must be providing some capacity of informal (unpaid) care for a patient meeting patient eligibility criteria. If a patient unexpectedly becomes deceased during the study period, caregivers will be allowed to continue participation in the assigned study arm and complete study assessments if they wish to.
* Greater than or equal to 18 years of age.
* Ability to access study materials by internet or complete study activities in person as institutional and government policies allow.

Eligible patients include those who:

* Have new or recurrent American Joint Committee on Cancer (AJCC) stage I-IV head and neck cancer.
* Are receiving cancer treatment or awaiting planned treatment initiation, excluding those receiving neoadjuvant surgery or surgery only.
* Patients must be ambulatory and up more than 50% of waking hours, as measured by an ECOG Performance Status rating of level 0, 1, or 2.
* Greater than or equal to 18 years of age.
* Ability to access study materials by internet or complete study activities in person as institutional and government policies allow.
* Patients must be receiving some capacity of informal care from a caregiver meeting the above criteria. If the caregiver unexpectedly becomes deceased during the study period, the patient will be un-enrolled from this study as we are evaluating a caregiver-only delivered intervention.

Exclusion Criteria:

Caregivers will be excluded if:

• Cannot read/communicate in English

Patients will be excluded if they:

• Cannot read/communicate in English

Eligibility to participate in the study is conditional on participation of both the caregiver and patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandylen Nightingale, PhD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CONNECT Intervention Group - Group A | CONNECT Comparison Group - Group B
Started | 18 | 22
Completed | 18 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CONNECT Intervention Group - Group A | CONNECT Comparison Group - Group B | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Customized [Count of Participants; unit: Participants]
  Age 18-35 | 1 | 0 | 1
  Age 36-54 | 1 | 1 | 2
  Age 55-72 | 5 | 3 | 8
  Age unknown | 11 | 18 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 15 | 19 | 34
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 22 | 40
Some College Education [Count of Participants; unit: Participants] | 12 | 16 | 28
Married/ Partnered to Patient [Count of Participants; unit: Participants] | 12 | 16 | 28
Adult Children to Patient [Count of Participants; unit: Participants] | 5 | 2 | 7
Partnered. Married [Count of Participants; unit: Participants] | 13 | 19 | 32

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Caregivers Who Agree to Participate
Description: Number of caregivers who agreed to participate divided by the number of months of recruitment
Time Frame: 19 months
Population: The 40 participants that agreed to participate in the intervention were accrued over a total of 19 months.
Measure: Number; unit: participants per month
Groups:
- Accrual: Total number of caregivers that agreed to participate divided by the number of months of recruitment.
Arm/Group | Accrual
Number analyzed (Participants) | 40
participants per month | 2.1

2. Primary Outcome: Number of Eligible Participants
Description: Number of eligible participants who agreed to participate
Time Frame: 9 months
Population: Out of 108 participants found to be eligible to participate in the study intervention only 40 agreed and consented to begin the study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Participation: Number of screened participants found to be eligible versus participants who agreed to participate
Arm/Group | Participation
Number analyzed (Participants) | 108
Participants | 40

3. Primary Outcome: Number of Retention of Participants
Description: Number of participants who completed the T2 assessment divided by the number who agreed to participate
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Retention: Number of participants who completed the assessment divided by the number who agreed to participate
Arm/Group | Retention
Number analyzed (Participants) | 40
Participants | 32

4. Primary Outcome: Acceptability - (Intervention Arm Only)
Description: Survey developed for study to assess how much caregivers liked different aspects of CONNECT; and a ~30min (approximately) qualitative interview to further explore acceptability (measures were not at all helpful, a little helpful, somewhat helpful or quite a bit helpful).
Time Frame: 9 months
Population: The acceptability measures were obtained from only 1 arm (intervention arm, since the questions pertain to the acceptability of the intervention), and were asked at the final time point, which means the n is those left in the intervention arm at the last time point.
Measure: Count of Participants; unit: Participants
Groups:
- Acceptability (Intervention Arm Only): Survey developed for study to assess how much caregivers liked different aspects of CONNECT; and a ~30min (approximately) qualitative interview to further explore acceptability.
Arm/Group | Acceptability (Intervention Arm Only)
Number analyzed (Participants) | 12
Participants
  Educational video on the CONNECT website (step 1 in guide): Not at all helpful | 1
  Educational video on the CONNECT website (step 1 in guide): A little helpful | 3
  Educational video on the CONNECT website (step 1 in guide): Somewhat helpful | 5
  Educational video on the CONNECT website (step 1 in guide): Quite a bit helpful | 3
  Online survey to identify the types of resources/services that might be helpful as a caregiver: Not at all helpful | 2
  Online survey to identify the types of resources/services that might be helpful as a caregiver: A little helpful | 2
  Online survey to identify the types of resources/services that might be helpful as a caregiver: Somewhat helpful | 4
  Online survey to identify the types of resources/services that might be helpful as a caregiver: Quite a bit helpful | 4
  List of supportive care resources: Not at all helpful | 2
  List of supportive care resources: A little helpful | 2
  List of supportive care resources: Somewhat helpful | 5
  List of supportive care resources: Quite a bit helpful | 3
  Referral option immediately upon completing the survey to identify resource interest: Not at all helpful | 1
  Referral option immediately upon completing the survey to identify resource interest: A little helpful | 2
  Referral option immediately upon completing the survey to identify resource interest: Somewhat helpful | 7
  Referral option immediately upon completing the survey to identify resource interest: Quite a bit helpful | 2
  2 week follow up phone call to discuss available resources: number analyzed (Participants) | 10
  2 week follow up phone call to discuss available resources: Not at all helpful | 1
  2 week follow up phone call to discuss available resources: A little helpful | 2
  2 week follow up phone call to discuss available resources: Somewhat helpful | 6
  2 week follow up phone call to discuss available resources: Quite a bit helpful | 1

5. Primary Outcome: Acceptability - (Intervention Arm Only)
Description: Survey developed for study to assess how much caregivers liked different aspects of CONNECT; and a ~30min (approximately) qualitative interview to further explore acceptability (measures were strongly agree, agree and undecided).
Time Frame: 9 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Acceptability (Intervention Arm Only)
Number analyzed (Participants) | 14
Participants
  Strongly Agree | 2
  Agree | 7
  Undecided | 5

6. Other Pre Specified Outcome: SF-12 Patient Measures - Physical/Emotional Well-being
Description: A 12-item instrument measuring physical and mental well-being, though our analyses will focus on physical well-being; widely used in oncology populations. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: 1 year
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Unplanned Healthcare Utilization Survey
Description: Unplanned healthcare utilization survey will be calculated using a one item continuous score. The survey will capture patient self-reported unplanned healthcare utilization (number of unplanned visits to the emergency room, urgent care, or healthcare provider) from time points of baseline to end of treatment.
Time Frame: 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: FAMCARE Questionnaire (Patient)
Description: A 20-item instrument with 4 subscales to assess family caregiver satisfaction with information giving, availability of care, physical patient care, and symptom control. Participants will answer questions to indicate how satisfied they are with care family member has received. (Subscales = (S) satisfied, (U) undecided, (D) dissatisfied or (VD) very dissatisfied
Time Frame: 1 year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: PROMIS Emotional Distress-Anxiety-Short Form 8a for Patients
Description: An 8-item instrument that assesses fear, anxious misery, hyperarousal, and somatic symptoms related to arousal; widely used in oncology populations
Time Frame: 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: PROMIS Emotional Distress- Depression-Short Form 8a for Patients
Description: An 8-item instrument that assesses sadness, guilt, self-criticism, worthlessness, loneliness, interpersonal alienation, as well as loss of interest, meaning, and purpose.Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of anxiety.
Time Frame: 1 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Patient - Quality of Life Functional Assessment of Cancer Therapy - Head and Neck (FACT-H&N)
Description: A 39-item instrument that measures physical, social, emotional, and functional well-being, as well as additional head and neck-related concerns. Scoring scale is 0 = not at all to 4 = very much). Maximum score of 156. Higher scores indicate a better quality of life.
Time Frame: 1 year
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Supportive Care Utilization
Description: Adapted version of the 28-item Consumer-Based Cancer Care Value Index- Services and Resources instrument assessing use of services to meet multidimensional supportive needs. Intervention caregivers will also self-report service use by completing an auto-generated REDCap survey to query about utilization of the specific resources that each caregiver expressed interest in accessing.
Time Frame: 1 year
Reporting Status: Not Posted

13. Other Pre Specified Outcome: FAMCARE Questionnaire (Caregiver)
Description: as for outcome 8
Time Frame: 1 year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Caregiver Reaction Assessment
Description: Caregiver Reaction Assessment - 24-item instrument assessing positive and negative aspects of caregiving (esteem, lack of family support, finances, schedule, and health). The CRA has been tested in cancer caregivers; demonstrated validity and reliability. Each item is rated on a 1 to 4 scale. 1 (not at all) 2 (somewhat) 3 (quite a bit) 4 (completely)
Time Frame: 1 year
Reporting Status: Not Posted

15. Other Pre Specified Outcome: PROMIS Emotional Distress-Anxiety-Short Form 8a
Description: An 8-item instrument that assesses fear, anxious misery, hyperarousal, and somatic symptoms related to arousal; widely used in oncology populations. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of anxiety.
Time Frame: 1 year
Reporting Status: Not Posted

16. Other Pre Specified Outcome: PROMIS Emotional Distress- Depression-Short Form 8a
Description: An 8-item instrument that assesses sadness, guilt, self-criticism, worthlessness, loneliness, interpersonal alienation, as well as loss of interest, meaning, and purpose. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression.
Time Frame: 1 year
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Caregiver Quality of Life Index-Cancer (CqoL-Canc)
Description: 35-item instrument assessing dimensions of caregiver quality of life (burden, disruptiveness, positive adaptation, financial concerns). Scoring scale is 0 = not at all to 4 = very much). Maximum score of 140. Higher scores indicate better quality of life.
Time Frame: 1 year
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Caregiver Risk Scale
Description: A 7-item measure to assess caregiver behaviors for managing self-care. Questions are answered Yes or No and is a summation of the number of risks. Score range of 0-7, the higher the number, the greater the risk.
Time Frame: 1 year
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Caregiver Adherence to Referral Survey
Description: Survey responses will be coded as "adhered" or "did not adhere" for agency- and caregiver- reported service utilization. The score reporting is a dichotomous outcome of an adhered or not adhered.
Time Frame: 1 year
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Caregiving Self-Efficacy Scale
Description: 21-item instrument assessing caregivers' perceived self-efficacy for coping with cancer (managing medical information, caring for care recipient, caring for oneself, managing difficult interactions/emotions). Uses a likert scale from 1 (not at all confident) to 9 (totally confident). Higher scores indicate higher self-efficacy for coping with cancer.
Time Frame: 1 year
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Barriers to Supportive Care Use Survey
Description: A 16-item survey with an additional "other" category for a caregiver to report additional barriers not noted on the survey. Response options range from never (0) to always (4). Higher scores indicate a greater number of barriers.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | CONNECT Intervention Group - Group A | CONNECT Comparison Group - Group B
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03875885/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT03875885/ICF_001.pdf